CLINICAL TRIAL: NCT05613439
Title: The Fast-track Centre for Hip and Knee Replacement Prospective Database on Preoperative Patientcharacteristics and Postoperative Complications
Brief Title: The Fast-track Centre for Hip and Knee Replacement Database
Acronym: FCD
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other); Gødstrup Hospital (Other); Sygehus Lillebaelt (Other); Svendborg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Naestved Hospital (Other); Bispebjerg Hospital (Other); Aalborg University Hospital (Other); Hvidovre University Hospital (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christoffer Joergensen, Database manager, Rigshospitalet, Denmark
Other Study IDs: FC-1
Record Dates: First submitted 2022-10-19; First posted 2022-11-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hip; Knee; Fast-track Surgery; Enhanced Recovery After Surgery; Perioperative Medicine; Ambulatory Surgical Procedures; Perioperative/Postoperative Complications; Patient Satisfaction
Keywords: Hip Replacement; Knee Replacement; Perioperative Medicine; Enhanced Recovery After Surgery; Perioperative/Postoperative Complications; Ambulatory Surgical Procedures
MeSH Terms: conditions — Postoperative Complications; Patient Satisfaction | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Day-surgery group: Patients having hip or knee replacement as day-surgery with successful discharge to own home on day of surgery
  Interventions: Procedure: Day-surgery
- High-risk patients: Patients evaluated to be at increased risk of postoperative complications. These patients will receive relevant additional attention based on type of comorbidity. I.e. preoperative evaluation of iron status and i.v. iron treatment in case of preoperative anaemia, increased focus on avoidance of NSAIDs and adequate fluid therapy in patients with renal disease etc.
  Interventions: Procedure: High-risk patient
- Main group: Patients who are not scheduled for day-surgery and without comorbidities qualifying as "high-risk". These patients go through a standard fast-track procedure with discharge to own home when fulfilling functional discharge criteria.
  Interventions: Procedure: Main Group

INTERVENTIONS:
Procedure: Day-surgery — Standard surgical procedure but with planned discharge on day of surgery
  Groups: Day-surgery group
Procedure: High-risk patient — Standard fast-track procedure but with additional perioperative measures dependent on risk-profile.
  Groups: High-risk patients
Procedure: Main Group — Standard fast-track procedure according to usual standard of care and discharge when fulfilling functional discharge criteria
  Groups: Main group

SUMMARY:
This is a prospective study-registry on preoperative patient characteristics and postoperative complications in patients having fast-track hip and knee replacement surgery in 8 Danish dedicated arthroplasty departments from all five health regions in Denmark. The registry consists of detailed patient and physician reported preoperative characteristics and including prescribed medication and lab results. Follow-up is based on electronical medical records by dedicated nurses with physician backup and includes Clavien-Dindo and Comprehensive Complication Index scoring. All patients having day-surgery also completes a patient reported questionaire on health-care utilization and return to work by day 30. Finally, a machine-learning algorithm for identification of "high-risk" patients based on he preoperative data is included.

DETAILED DESCRIPTION:
The study registry is intended for further detailed research on postoperative morbidity, feasibility and safety of day surgery and functional outcomes after fast-track hip and knee replacement in 8 dedicated Danish arthroplasty wards across all five health care regions in Denmark. The work is a continuation of the Lundbeck Foundation Centre Database on Hip and Knee Replacement also registered in ClinicalTrials but ceased enrolling in august 2017.

The aim of the registry is to provide standardized and comprehensive information on preoperative patient characteristics and postoperative complications, patient reported outcome measures and health-care utilization in fast-track hip and knee replacement within a socialized health-care system. Each department have dedicated research personel assuring registration and follow-up supervised by a datamanager, and with database-support from the Danish health Region of Southern Denmark.

All departments have similar established fast-track protocols as standard of care, but with focus on dividing patients into day-surgery, main fast-track group and high-risk cohorts.

Preoperative data includes information on prescribed medication, Clinical Frailty Score using CFS v.1, evaluation of Pain Catastrophizing Scale as well as laboratory testing of hemoglobin, kidney function, Hb1Ac in diabetics and C-reactive protein level. On the basis of the collected preoperative data a machine-learning algorithm for identifying the "high-risk" patients is being refined and with planned induction in the database.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* non-malignant surgery
* danish social security number
* elective procedure

Exclusion Criteria:

* unwilling to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participating dedicated arthroplasty departments are placed in either large university or regional hospitals. The departments cover all five healthcare regions in Denmark and are estimated to contribute with about 40% of the annual hip and knee replacements in Denmark. Thus, the population is representative of the general Danish arthroplasty population.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fraction of unselected patients able to undergo day-surgery procedures | 7 days postoperatively
  The fraction patients eligible for day-surgery who are discharged on day of surgery.
postoperative morbidity | 90 days postoperatively
  postoperative morbidity resulting in prolonged (>2 days) hospitalisation, readmissions or mortality 90 days after surgery.
postoperative morbidity Clavien-Dindo | 90 days postoperatively
  Postoperative morbidity resulting in prolonged (>2 days) hospitalisation, readmissions or mortality 90 days after surgery according to the Clavien-Dindo index.
postoperative morbidity CCI | 90 days postoperatively
  Postoperative morbidity resulting in prolonged (>2 days) hospitalisation, readmissions or mortality 90 days after surgery according to the Comprehensive Complication Index

SECONDARY OUTCOMES:
Healthcare utilisation in day-surgery | 30 days postoperatively
  Registration of emergency room visits, visits to general practitioners and use of medical emergency services within 30 days after having hip or knee replacement as day-surgery procedure.

OTHER OUTCOMES:
return to work in day-surgery | 30 days postoperatively
  changes in work status and time to return to work in day-surgery procedures
patient satisfaction and patient reported outcome measures1 | Baseline, 90 and 365 days postoperatively
  collection of data on patient satisfaction and function after surgery using the EQ-5D-5L (score from 0-100 with increasing score indicating better health)
patient satisfaction and patient reported outcome measures, THA only. | Baseline, 90 and 365 days postoperatively
  collection of data on patient satisfaction and function after surgery using the Oxford Hip Score (range from 0-48 with increasing score indicating better function).
patient satisfaction and patient reported outcome measures, TKA only. | Baseline, 90 and 365 days postoperatively
  collection of data on patient satisfaction and function after surgery using the Oxford Knee score (range from 0-48 with increasing score indicating better function).

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, M.D., Study Chair — Section for Surgical Pathophysiology, Rigshospitalet, University of Copenhagen
Locations (8):
- Denmark (8):
  - Bispebjerg University Hospital, Copenhagen, Capital Region
  - Gentofte University Hospital, Gentofte Municipality, Capital Region
  - Hvidovre Hospital, Hvidovre, Capital Region
  - Gødstrup Hospital, Herning, Region of Middle Judland
  - Aalborg University Hospital, Farsø, Farsø, Region of Northern Judland
  - Lillebaelt Hospital, Vejle, Vejle, Region of Sourthern Denmark
  - Næstved Hospital, Næstved, Region Sjælland
  - University Hospital Svendborg, Svendborg, Region Syddanmark

REFERENCES:
- [Derived] Issa LM, Jorgensen CC, Madsbad S, Lindberg-Larsen M, Varnum C, Jakobsen T, Andersen MR, Bieder MJ, Overgaard S, Hansen TB, Gromov K, Kehlet H. Feasibility of a prospective multicenter observational study-is diabetes a risk factor in ERAS joint arthroplasty? Pilot Feasibility Stud. 2025 Dec 13. doi: 10.1186/s40814-025-01747-w. Online ahead of print. PMID 41387916
- [Derived] Mahmoud LI, Kehlet H, Madsbad S, Lindberg-Larsen M, Varnum C, Jakobsen T, Andersen MR, Bieder MJ, Overgaard S, Hansen TB, Gromov K, Jorgensen CC. Perioperative GLP1-RA management and risk of aspiration in patients with diabetes undergoing fast-track hip and knee arthroplasty. Dan Med J. 2025 Apr 9;72(5):A09240629. doi: 10.61409/A09240629. PMID 40407287
- [Derived] Jorgensen CC, Lindberg-Larsen M, Gromov K, Varnum C, Bider MJ, Overgaard S, Andersen MR, Hansen TB, Kehlet H. Association of non-anaemic iron deficiency with postoperative outcomes after fast-track hip and knee arthroplasty: a prospective cohort study. Br J Anaesth. 2025 Aug;135(2):322-330. doi: 10.1016/j.bja.2025.03.039. Epub 2025 May 21. PMID 40404500
- [Derived] Issa LM, Kehlet H, Madsbad S, Lindberg-Larsen M, Varnum C, Jakobsen T, Andersen MR, Bieder MJ, Overgaard S, Hansen TB, Gromov K, Jorgensen CC. Protocol for a prospective multicentre cohort study to address the question whether diabetes and its management is still a risk factor in fast-track joint arthroplasty. BMJ Open. 2024 Apr 23;14(4):e080232. doi: 10.1136/bmjopen-2023-080232. PMID 38658012
- See also: The Fast-track Center Homepage — https://fast-track.health/